CLINICAL TRIAL: NCT06042751
Title: Randomized Comparison of a Telemedicine-supported Psychosomatic Intervention, a Physical Activity Intervention and the Combination of Both in Patients With Post-covid19 Syndrom.
Brief Title: Psychosomatic, Physical Activity or Both for Post-covid19 Syndrom
Acronym: TELPOCO
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hannover Medical School (Other)
Collaborators: Health Insurance Audi BKK (Unknown); occupational health service Volkswagen AG (Unknown); Helmholtz Centre for Infection Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 9LZF23
Record Dates: First submitted 2023-09-05; First posted 2023-09-21 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Post-COVID-19 Syndrome
Keywords: Physical actvity; Psychotherapy; Cobined exercise and psychotherapy; Covid-19; Post-Covid-19-Syndrom
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; COVID-19 | interventions — Exercise Therapy; Psychotherapy

STUDY DESIGN:
Intervention Model Description: One study arm will receive exercise therapy with 6 treatments over three months.
  One study arm receives psychotherapy with 6 treatments over three months. One study arm receives combined exercise and psychotherapy over three months.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Exercise Therapy (Experimental): Six online consultations focusing on exercise therapy, each lasting 50 minutes every two weeks, resulting in 300 min in 3 months.
  Interventions: Behavioral: Exercise Therapy
- Psychotherapy (Experimental): Six online consultations focusing on psychotherapy, each lasting 50 minutes every two weeks, resulting in 300 min in 3 months.
  Interventions: Behavioral: Psychotherapy
- Combined exercise and psychotherapy (Experimental): Both interventions (exercise and psychotherapy) are combined. Six biweekly online session with 50% exercise therapy (a 25 min) and 50% psychotherapy (a 25 min) will take place, resulting in 300 min overall therapy in 3 months. The content of the procedure is simultaneous to the interventions described in the exercise therapy arm and the psychotherapy arm, respectively.
  Interventions: Behavioral: Exercise Therapy; Behavioral: Psychotherapy

INTERVENTIONS:
Behavioral: Exercise Therapy — Six online consultations will take place on the basis of the sports medicine assessment every two weeks, resulting in 300 min in 3 months. For the home-based implementation, participants receive wearables with which the activity and training data are collected. In conjunction with feedback, the goal is to ensure that the interventions lead to improvements in self-control, reduced resilience, and fatigue without overwhelming participants with volume or intensity. Due to the expected large differences in personal performance, determined in the initial assessment, the exercise plan is individually designed and regularly adjusted. This includes control of everyday activity as well as moderate endurance and strengthening exercises totalling up to 30min daily. The individual training intensity is below the aerobic lactate threshold so that overload is avoided. The average training heart rate is planned to be in the range between 50 and 70% of the maximum heart rate.
  Arms: Combined exercise and psychotherapy; Exercise Therapy
Behavioral: Psychotherapy — Six online consultations will take place based on the psychosocial assessment and the initial psychosomatic interview every two weeks, resulting in 300 min in 3 months. A structured, telemedicine-supported, modularized, brief psychosomatic intervention is planned with a focus on psychoeducational elements, promotion of self-management, improvement of illness acceptance, modification of self-monitoring, and learning to cope with altered performance levels. The six modularized telemedical sessions taking into account the specific deficits identified in the psychosomatic evaluation. Within the sessions, starting points are identified with the patients, which the patients can work on independently between the sessions.
  Arms: Combined exercise and psychotherapy; Psychotherapy

SUMMARY:
Post-Covid(PoC)-patients with fatigue symptoms respond very differently to physical rehabilitation programs. While PoC-patients with psychological symptoms benefit little from physical interventions, fatigue and exercise capacity improves significantly without the presence of psychological symptoms. RCT studies on effects of psychotherapy or the combination of phsical activity with psychotherapy in PoC are not yet available. Therefore, the aim is to investigate the unimodal effects of psychotherapy and exercise therapy or the combination of both on fatigue in PoC patients with fatigue in a randomized clinical trial. Patients will be assigned to the three intervention groups (psychotherapy, physical rehabilitation, combination of both) stratified for sex, gender and BMI status.

The intervention duration is 3 months with therapeutic online sessions for 50 min every 2 weeks. After another 3 months without intervention, the sustainability will evaluated. Secondarily, the investigators analyzes which patient benefits most from which therapeutic approach and seek for specific predictors of patient´s individual response.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged over 18 and
* diagnosed post-Covid-19 syndrome: (positive PCR or antibody test) and Fatigue Assessment Scale (FAS) ≥ 22 points

Exclusion Criteria:

* Current participation in another intervention study
* Illnesses or functional disorders that potentially explain the fatigue symptoms otherwise
* Any illness or impairment that the examining physician judges to preclude participation in a physical training intervention
* Suicidality or severe mental illness (e.g. mania, acute phase of schizophrenia) that requires acute treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 195 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Fatigue | The questionnaire will be completed at baseline, after the intervention (after 3 months), and after another 3-month observation period (after 6 months).
  Measured with the Fatigue Assessment Scale (FAS). The FAS is a 10-question assessement scale with five questions related to physical fatigue and 5 questions (questions 3 and 6-9) related to mental fatigue. The total score ranges from 10 to 50. A total FAS score < 22 indicates no fatigue, a score ≥ 22 indicates fatigue, and a score > 35 indicates extreme fatigue.

SECONDARY OUTCOMES:
Health-related quality of life | The questionnaire will be completed at baseline, after the intervention (after 3 months), and after another 3-month observation period (after 6 months).
  Measured with the Short Form-36 (SF-36) questionnaire. The 36 questions of the SF-36 are designed to reflect 8 domains of health, including physical functioning, physical role, pain, general health, vitality, social functioning, emotional role, and mental health. The range is 0-100, with higher scores indicating higher quality of life. In addition, a physical (PCS) and mental (MCS) composite score can be calculated.
Depression and Anxiety | The questionnaire will be completed at baseline, after the intervention (after 3 months), and after another 3-month observation period (after 6 months).
  Measured with the Hospital Anxiety and Depression Scale (HADS). The HADS questionaire consists of fourteen items pertaining to the two subscales for anxiety and depression. Scores for the anxiety and depression subscale range from 0 to 21, with higher score indicating more severe anxiety or depression. Values can be interpreted as normal from 0-7 points, mild (8-10 points), moderate (11-14 points), and severe (15-21 points).
Physical and psychological fatigue severity | The questionnaire will be completed at baseline, after the intervention (after 3 months), and after another 3-month observation period (after 6 months).
  Measured with the Chalder Fatigue Skala (CFS). The 11-part self-report instrument consists of a total scale and two subscales, physical and psychological fatigue. The maximum total score is 33, with higher scores indicating higher levels of fatigue. The maximum score for physical fatigue is 21 (7 items) and for mental fatigue is 12 (4 items). Additionally, a binary code can be calculated for each of the 11 items (0 and 1 = 0; 2 and 3 = 1) to identify cases of severe fatigue. A total score of 4 or more indicates severe fatigue.
Post-exertional malaise | The questionnaire will be completed at baseline, after the intervention (after 3 months), and after another 3-month observation period (after 6 months).
  The post-exertional malaise scale (PEM-scale) uses five different 5-point Likert scales to assess the frequency or severity of PEM symptoms and a 7-point Likert scale to assess the duration of PEM evaluate resulting in a maximum score of 46.
Multidimensional Fatigue Inventory | The questionnaire will be completed at baseline, after the intervention (after 3 months), and after another 3-month observation period (after 6 months).
  The Multidimensional Fatigue Inventory questionaire (MFI-20) is a 20-item self-assessment instrument consisting of five subscales: (1) general fatigue, (2) physical fatigue, (3) decreased activity, (4) decreased motivation, and (5) mental fatigue. Each subscale consists of four items with response options on a five-point Likert scale (1 = yes, that applies, 5 = no, that does not apply). Higher scores indicate higher levels of fatigue
Disability | The questionnaire will be completed at baseline, after the intervention (after 3 months), and after another 3-month observation period (after 6 months).
  The Bell Disability Scale includes eleven statements about the level of physical function. The scale is rated in increments of 10, from 0 (very severe, constantly bedridden) to 100 (healthy).
Work ability | The questionnaire will be completed at baseline, after the intervention (after 3 months), and after another 3-month observation period (after 6 months).
  The work ability index questionnaire (WAI) contains seven questions concerning work, work ability and health, resulting in a total score ranging from seven to 49, with higher values representing greater work ability.
Illness Perception | The questionnaire will be completed at baseline, after the intervention (after 3 months), and after another 3-month observation period (after 6 months).
  The Brief Illness Perception Questionnaire (IPQ) assesses cognitive and emotional illness perception. The here used short IPQ contains eight new items as well as part of the causal scale previously used in the IPQ-R. All items except the causal question are rated on a scale of 0 to 10. Five of the items assess cognitive representations of illness: consequences (Item 1), time frame (Item 2), personal control (Item 3), treatment control (Item 4), and identity (Item 5). Two of the items capture emotional representations: concern (item 6) and feelings (item 8). One item assesses the comprehensibility of the illness (Item 7). The causal representation is assessed using an open-response item in which patients are asked to list the three most important causal factors for their illness (Item 9)

CONTACTS AND LOCATIONS:
Overall Officials: Uwe Tegtbur, Principal Investigator — Hannover Medical School, Institute for Sports Medicine
Locations (1):
- Hannover Medical School, Hanover, Lower Saxony, Germany

REFERENCES:
- [Derived] Beyer S, Nohre M, Pink I, Hackl S, Thomas NH, Klawonn F, Tegtbur U, de Zwaan M, Haufe S. Comparison of telemedicine-assisted psychotherapy, exercise therapy, or a combination of both in patients with post-COVID-19 syndrome (TelPoCo): study protocol for a randomized controlled trial. Trials. 2025 Jul 20;26(1):251. doi: 10.1186/s13063-025-08968-7. PMID 40685367